CLINICAL TRIAL: NCT03118193
Title: Biomarkers of Antidepressant Resistance - BIORESA
Brief Title: Biomarkers of Antidepressant Resistance
Acronym: BIORESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHAO16-WEH/BIORESA
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: depression; antidepressant; resistance
MeSH Terms: conditions — Depression | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Depressive patient (Experimental): olfactive tests ; blood test ; optional: Tissue Pulsatility imaging ; optional: Collection of faeces
  Interventions: Other: olfactive tests; Biological: blood test; Biological: Collection of faeces; Device: Tissue Pulsatility imaging

INTERVENTIONS:
Other: olfactive tests — olfactive tests: odor identification, odor discrimination and olfactory threshold
Biological: blood test — one sample of 4mL
Biological: Collection of faeces — Collection of faeces by patient at home - optional
Device: Tissue Pulsatility imaging — Ultrasound exploration of brain pulsatility - optional

SUMMARY:
According to the WHO, major depressive disorders have become the second worldwide cause of disability. Treatment, long-term medication, leads to frequent resistance (up to 40%).

Establishing a cerebral molecular signature of depression is not feasible in humans (need for cerebral samples). The alternative is to use peripheral biological samples (blood, urine, saliva).

Metabolomic is the integrated and quantitative study of all the metabolites of a biological system. This aims to define the metabolic status of an organism for a particular condition.

Metabolites are derived from biological extracts (cells, tissues, serum, plasma, urine, etc.) and are detected by:

* liquid or gas chromatography coupled to mass spectrometry (LC-MS, GC-MS),
* proton nuclear magnetic resonance (1 H-NMR). The biomarkers resulting from these studies have become important diagnostic criteria, measured objectively and evaluated as indicators of a normal or pathological state, or even predictors of treatment efficacy.

This approach allows the discovery of biomarkers that best describe the status of a disease for better understanding and are usable in a context of individualized medicine, with effects on clinical practice and management.

ELIGIBILITY:
Inclusion Criteria:

* between 18-60 years-old
* major depressive disorder, confirmed by Mini International Neuropsychiatric Interview (MINI)
* no bipolar disorder or schizophrenia, confirmed by MINI
* no neurological dementia disease
* able to perform olfactive tests, i.e. no anosmia and/or allergy to odors
* score MADRS (Montgomery AsbergDepression Rating Scale) >20
* no antidepressant treatment during 14 days before inclusion
* informed written consent
* affiliation to a social security system

Exclusion Criteria:

* patient who don't want any antidepressant treatment for this depressive episode
* legal incapacity and/or any circumstances making the person unable to understand the trial features, purposes or consequences
* participating to drug clinical study or in exclusion period of clinical study because of previous participation
* pregnant woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
metabolic print of blood | 2 months
  Metabolome of blood

SECONDARY OUTCOMES:
olfactive identification | 2 months
  Olfactive response: odor identification
olfactive discrimination | 2 months
  Olfactive response: odor discrimination
Olfactory threshold | 2 months
  Olfactive response: olfactory threshold
Microbiote of faeces | 2 months
  Bacteria of faeces
Maximal measures of brain pulsatility | 2 months
  Maximal brain pulsatility
Mean measures of brain pulsatility | 2 months
  Mean brain pulsatility
Metabolic print of faces | 2 months
  Metabolome of faeces

CONTACTS AND LOCATIONS:
Overall Officials: Wissam El-Hage, PhD, Principal Investigator — CHRU TOURS
Locations (1):
- CHU Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Desmidt T, Dujardin PA, Brizard B, Remenieras JP, Gissot V, Dufour-Rainfray D, Atanasova B, Kazour F, Belzung C, Camus V, El-Hage W. Decrease in ultrasound Brain Tissue Pulsations as a potential surrogate marker of response to antidepressant. J Psychiatr Res. 2022 Feb;146:186-191. doi: 10.1016/j.jpsychires.2021.12.056. Epub 2022 Jan 3. PMID 34995994